CLINICAL TRIAL: NCT03537573
Title: Provider-Targeted Behavioral Interventions to Prevent Unsafe Opioid Prescribing for Acute Non-Cancer Pain in Primary Care
Brief Title: Provider-Targeted Behavioral Interventions to Prevent Unsafe Opioid Prescribing for Acute Pain in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Geisinger Clinic (Other); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20110336; UOP-1609-36881 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2018-04-29; First posted 2018-05-25 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-06

CONDITIONS: Acute Pain; Headache; Musculoskeletal Pain
Keywords: Pragmatic clinical trial; Primary care; Provider-targeted; Behavioral intervention; Electronic health record
MeSH Terms: conditions — Acute Pain; Headache; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: 48 primary care clinics (N=19,855 patients participants anticipated) randomized to 4 arms in 2x2 factorial design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care/Guideline (Active Comparator): The Usual Care group (also known as the Guideline group) follows the recent Center for Disease Control (CDC) guidelines and, when triggered by an opioid prescription during a qualifying visit, will be delivered real-time in a short checklist of recommendations to: 1) check the state-specific Prescription Drug Monitoring Program; 2) assess risk factors for opioid-related harms (e.g., history of substance use disorder, history of mental health problems, benzodiazepine use); 3) avoid extended-release or long-acting opioids; 4) use a low dose of immediate-release opioid for short period of time (3-7 days); and 5) consider non-opioid management such as acetaminophen, non-steroidal anti-inflammatory agents (NSAIDS), and physical therapy. Epic EHR order sets will be linked to enable easing ordering of non-opioid therapy.
  Interventions: Behavioral: Usual Care/Guideline
- Guideline + Opioid Justification (OJ) (Experimental): Providers will be required asked to enter a free text justification for their decision to prescribe an opioid analgesic for the acute pain condition. The provider will be notified that the justification provided will be visible in the Epic EHR. The provider has the option of entering a justification or not. If no justification is entered, nothing will be entered into the record (i.e., the Opioid Justification area in the encounter record will be left blank). The provider does not need to enter a justification if they choose to cancel the opioid prescription.
  Interventions: Behavioral: Usual Care/Guideline; Behavioral: Opioid Justification
- Guideline + Provider Comparison (PC) (Experimental): Providers will receive monthly feedback via e-mail on their status in regards to initial opioid prescriptions for acute pain, adherence to safe opioid prescribing guidelines, and proportion of patients started on opioids f or acute pain who transition to chronic opioid therapy (> 3 months). Providers in the lowest decile overall for proportion of patients with initial opioid prescriptions , unsafe opioid prescribing, and transition to chronic opioid therapy (> 3 months) will be given positive feedback for providing high quality, evidence-based care to their patients with acute pain. Providers outside the lowest decile will be notified they are outside the high quality, evidence-based care range and will be provided with their proportions compared to the high performers.
  Interventions: Behavioral: Usual Care/Guideline; Behavioral: Provider Comparison
- Guideline + OJ + PC (Experimental): This arm will include the guideline, opioid justification, and provider comparison described above.
  Interventions: Behavioral: Usual Care/Guideline; Behavioral: Opioid Justification; Behavioral: Provider Comparison

INTERVENTIONS:
Behavioral: Usual Care/Guideline — The Usual Care group (also known as the Guideline group) follows the recent CDC guidelines and, when triggered by an opioid prescription during a qualifying visit, will be delivered real-time in a short checklist of recommendations to: 1) check the state-specific Prescription Drug Monitoring Program; 2) assess risk factors for opioid-related harms (e.g., history of substance use disorder, history of mental health problems, benzodiazepine use); 3) avoid extended-release or long-acting opioids; 4) use a low dose of immediate-release opioid for short period of time (3-7 days); and 5) consider non-opioid management such as acetaminophen, non-steroidal anti-inflammatory agents (NSAIDS), and physical therapy. Epic EHR order sets will be linked to enable easing ordering of non-opioid therapy.
Behavioral: Opioid Justification — Providers will be required asked to enter a free text justification for their decision to prescribe an opioid analgesic for the acute pain condition. The provider will be notified that the justification provided will be visible in the Epic EHR. The provider has the option of entering a justification or not. If no justification is entered, nothing will be entered into the record (i.e., the Opioid Justification area in the encounter record will be left blank). The provider does not need to enter a justification if they choose to cancel the opioid prescription.
  Arms: Guideline + OJ + PC; Guideline + Opioid Justification (OJ)
Behavioral: Provider Comparison — Providers will receive monthly feedback via e-mail on their status in regards to initial opioid prescriptions for acute pain, adherence to safe opioid prescribing guidelines, and proportion of patients started on opioids or acute pain who transition to chronic opioid therapy (> 3 months). Providers in the lowest decile overall for proportion of patients with initial opioid prescriptions, unsafe opioid prescribing, and transition to chronic opioid therapy (> 3 months) will be given positive feedback for providing high quality, evidence-based care to their patients with acute pain. Providers outside the lowest decile will be notified they are outside the high quality, evidence-based care range and will be provided with their proportions compared to the high performers.
  Arms: Guideline + OJ + PC; Guideline + Provider Comparison (PC)

SUMMARY:
The investigators will assess whether behavioral science-based interventions can "nudge" providers towards more evidence-based care for patients with acute non-cancer pain.

Aim 1) Among opioid naïve primary care patients with acute non-cancer pain, compare the effect of the provider-targeted behavioral interventions (opioid justification and provider comparison), individually and in combination, on initial opioid prescription, initial use of non-opioid management, and patient-reported pain and function.

Aim 2) Compare the effect of the 2 provider-targeted behavioral interventions, individually and in combination, on unsafe opioid prescribing and transition to chronic opioid therapy.

Aim 3) Assess provider satisfaction and experience with the provider-targeted behavioral interventions.

Hypotheses:

Aim 1, H1a: Compared with the guideline (usual care) alone, the addition of the opioid justification and provider comparison behavioral interventions will be associated with a decreased proportion of opioid prescription and increased proportion of non-opioid management at the initial outpatient visit for acute non-cancer pain.

Aim 1, H1b: Compared with usual care (guideline) alone, the addition of the opioid justification and provider comparison behavioral interventions will be associated with no difference in patient-reported pain, function, and satisfaction at 1, 6, and 12 months.

Aim 2, H2: Compared with the usual care (guideline), the addition of opioid justification and provider comparison behavioral interventions will be associated with a decreased proportion of patients receiving unsafe opioid therapy and a decreased proportion of patients transitioning to chronic opioid therapy.

Study Design: Pragmatic, cluster-randomized clinical trial in 48 primary care clinics.

Study Population: The patient population will be 19,855 opioid naïve adults who present to clinic with acute uncomplicated musculoskeletal pain or headache.

Primary and Secondary Outcomes: The primary outcome measures will be receipt of an initial opioid prescription and unsafe opioid prescribing. Secondary outcomes will be non-opioid pain management, and, in 514 patients, patient-reported pain and function.

Analytic Plan: The investigators will test for differences in the primary and secondary outcomes among the 4 intervention groups.

Once completed, the project will provide evidence that health systems and other stakeholders need to implement interventions to prevent unsafe opioid prescribing.

ELIGIBILITY:
1. Patient Participants

   Inclusion Criteria:
   * Age 18 years or older; ii) index outpatient encounter with International Classification of Disease (ICD)-10 code for acute neck, back, or other musculoskeletal and headache diagnosis ("acute" defined as no similar diagnosis in past 3 months).

   Exclusion Criteria:
   * Cancer diagnosis (other than non-melanoma skin cancer)
   * Receipt of opioid prescription within 12 months of index outpatient encounter
2. Providers

Inclusion Criteria:

* Primary care provider (MD, Doctor of Osteopathy (DO), Physician Assistant (PA), Nurse Practitioner (NP)) at participating practice

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22616 (Actual)
Dates: Start 2018-09-23 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Initial Opioid Prescription | 1 day (assessed on day of initial qualifying clinic visit
  Initial opioid prescription (yes/no) (Primary) (Hypothesis 1a). Opioid prescription at qualifying clinic visit, measured via electronic health record (EHR).

SECONDARY OUTCOMES:
Initial non-opioid management | 1 day (assessed on day of initial qualifying clinic visit)
  Initial non-opioid management (yes/no) (Secondary) (Hypothesis 1a). Defined as order for any non-opioid management strategy at baseline (e.g., non-opioid medication, physical therapy, behavioral therapy), measured via EHR.
Change in Patient Reported Pain and Function | Assessed at 1, 6, and 12 months after initial qualifying clinic visit
  Change in Patient Reported Pain and Function (Secondary) (Hypothesis 1b). Measured by the 3-item Pain/Enjoyment/General Activities (PEG) instrument in clinic at baseline and via brief web survey or telephone interview
Unsafe opioid prescribing at 3 months | 3 months after initial qualifying clinic visit
  Defined over the prior 3 months as any of: a) receipt of initial extended release/long-acting opioid for acute pain; b) > 100 morphine milligram equivalent dose per day; c) opioid prescription in patients with substance use disorder or concurrent benzodiazepine prescription.
Unsafe opioid prescribing at 6 months | 6 months after initial qualifying clinic visit
  Defined over the prior 3 months as any of: a) receipt of initial extended release/long-acting opioid for acute pain; b) > 100 morphine milligram equivalent dose per day; c) opioid prescription in patients with substance use disorder or concurrent benzodiazepine prescription.
Unsafe opioid prescribing at 12 months | 12 months after initial qualifying clinic visit
  Defined over the prior 3 months as any of: a) receipt of initial extended release/long-acting opioid for acute pain; b) > 100 morphine milligram equivalent dose per day; c) opioid prescription in patients with substance use disorder or concurrent benzodiazepine prescription.
Chronic opioid therapy at 3 months | 3 months after initial qualifying clinic visit
  Chronic opioid therapy (Secondary) (Hypothesis 2). Ongoing, chronic opioid therapy will be measured via EHR
Chronic opioid therapy at 6 months | 6 months after initial qualifying clinic visit
  Chronic opioid therapy (Secondary) (Hypothesis 2). Ongoing, chronic opioid therapy will be measured via EHR
Chronic opioid therapy at 12 months | 12 months after initial qualifying clinic visit
  Chronic opioid therapy (Secondary) (Hypothesis 2). Ongoing, chronic opioid therapy will be measured via EHR

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L Kraemer, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Community Medicine Incorporated, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kraemer KL, Althouse AD, Salay M, Gordon AJ, Wright E, Anisman D, Cochran G, Fischer G, Gellad WF, Hamm M, Kern M, Wasan AD. Effect of Different Interventions to Help Primary Care Clinicians Avoid Unsafe Opioid Prescribing in Opioid-Naive Patients With Acute Noncancer Pain: A Cluster Randomized Clinical Trial. JAMA Health Forum. 2022 Jul 29;3(7):e222263. doi: 10.1001/jamahealthforum.2022.2263. eCollection 2022 Jul. PMID 35983579